CLINICAL TRIAL: NCT02655666
Title: Qingdao: Insulin Pump Follow-up Program
Status: Terminated | Type: Observational
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Other Study IDs: CEP303
Record Dates: First submitted 2015-12-18; First posted 2016-01-14 (Estimated); Results first posted 2018-09-21 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-04

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Medtronic MiniMed Paradigm® REAL-Time System: Medtronic MiniMed Paradigm® REAL-Time System consisting of Paradigm 722 Insulin Pump (MMT-722), Medtronic MiniLink® REAL-Time Transmitter (MMT-7703) and Sof-Sensor® (MMT-7003) Glucose Sensor

SUMMARY:
The purpose of the study is to observe/ collect clinical data, subject users' feedback, and device data to better understand the real-life usage and acceptance of the 722 Pump in type 1 diabetes subjects,<18 years of age, and the role of insulin pump therapy in Qingdao,China.

DETAILED DESCRIPTION:
This is a prospective, multi-center, non-randomized and noninterventional post-market release study. Subjects will participate in 2 phases with each phase requiring the subject to use the continuous subcutaneous insulin infusion (CSII) pump over the course of the study. During the study, subjects and parent or legal guardian will be trained to wear the glucose sensor in the abdominal area for 3 days to transmit real-time (RT) data to the pump. The duration of each study phase is approximately 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Subject is age < 18 years at time of screening
* Subject has a clinical diagnosis of type 1 diabetes
* Subject is willing to perform required sensor calibrations
* Subject is willing to wear the Medtronic MiniMed Paradigm® REAL Time System continuously throughout the study
* Subject is a participant in the Qingdao project.

Exclusion Criteria:

* Subject is actively participating in an investigational study (drug or device) wherein he/she has received diabetes treatment from an investigational study drug or investigational study devices in the last 2 weeks
* Subject has known hypersensitivity to insulin or insulin infusion set(including tape)
* Subject has used the insulin pump and/or real time CGM/sensor within 90 days before the screening visit for more than 10 days in the outpatient setting:

  * For example, subjects who have used insulin pump and/or real time CGM/sensor in the inpatient setting will still be eligible for enrollment.
  * For example, subjects who have used insulin pump and/or real time CGM/sensor for 8 days in the outpatient setting within 90 days before screening visit will still be eligible for enrollment.
  * For example, subjects who have worn the insulin pump and/or real time CGM/sensor for 3 months in the outpatient setting a year before the screening visit will still be eligible for enrollment
* Subject has been treated with drugs with a known effect on BG within 8 weeks before enrollment other than diabetes medications such as insulin or oral anti-diabetic agents.
* Subject has any systemic disease or medical condition found on screening that may interfere with the safety of the patient and efficacy of the study treatment, in the opinion of the Investigator, may preclude him/her from participating in the study.
* Subject is being treated for hyperthyroidism at time of screening
* Subject has taken any oral, injectable, or IV steroids within 8 weeks from time of screening visit, or plans to take any oral, injectable, or IV steroids during the course of the study
* Subject is currently abusing alcohol9. Any condition that either the Investigator believes would interfere with study participation or evaluation of results.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: A total of approximately 100 subjects (age<18 years) will be enrolled by up to 10 investigational centers to complete 13 scheduled study visits in the study.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2015-04; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tang Li, Principal Investigator — The Affiliated Hospital of Qingdao University; chunbin Wang, Principal Investigator — Chinese People's Liberation Army 401 Hospital; Yamie Zhu, Principal Investigator — Qingdao Endocrine and Diabetes Hospital
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Medtronic MiniMed Paradigm® REAL-Time System
Started | 16
Completed | 4
Not Completed | 12
Not completed — Sponsor stopped this clinical research. | 12

BASELINE CHARACTERISTICS:
Arm/Group | Medtronic MiniMed Paradigm® REAL-Time System
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.3 (2.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 5
Region of Enrollment [Number; unit: participants]
  China | 16

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated Hemoglobin (A1C)
Description: The change of A1C from baseline to end of study (1 year) will be presented
Time Frame: Change in A1C from baseline to end of study (1 year)
Population: Subject completed the study.
Measure: Mean (Standard Deviation); unit: percent Glycosylated Hemoglobin
Arm/Group | Medtronic MiniMed Paradigm® REAL-Time System
Number analyzed (Participants) | 4
percent Glycosylated Hemoglobin | 0.9 (2.22)

2. Secondary Outcome: Average Glucose Values Based on Continuous Glucose Monitoring Data
Description: The average glucose value of all available glucose value of each subject for each evaluation period is calculated, and we present the mean and std of the individual average glucose value for each evaluation period.
Time Frame: Data is collected during the 7 days following the end of each period (At end of month 3, no glucose data is collected).
Population: Subject enrolled with Continuous Glucose Monitoring (CGM) data available (Not all subjects have glucose value for analysis at each period.).
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Medtronic MiniMed Paradigm® REAL-Time System
Number analyzed (Participants) | 16
mmol/L
  Baseline: number analyzed (Participants) | 15
  Baseline | 9.8 (2.87)
  Month 6: number analyzed (Participants) | 12
  Month 6 | 10.4 (3.01)
  Month 9: number analyzed (Participants) | 6
  Month 9 | 9.5 (2.16)
  Month 12: number analyzed (Participants) | 3
  Month 12 | 8.0 (0.39)

3. Secondary Outcome: Standard Deviation of Glucose Value Based on Continuous Glucose Monitoring Data
Description: The standard deviation of all available glucose value of each subject for each evaluation period is calculated, and then we present the mean and std of the individual standard deviation for each evaluation period.
Time Frame: Data is collected 7 days following the end of each period (At end of month 3, no glucose data is collected.).
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Medtronic MiniMed Paradigm® REAL-Time System
Number analyzed (Participants) | 16
mmol/L
  Baseline: number analyzed (Participants) | 15
  Baseline | 3.5 (0.91)
  Month 6: number analyzed (Participants) | 12
  Month 6 | 3.0 (0.67)
  Month 9: number analyzed (Participants) | 6
  Month 9 | 3.0 (1.28)
  Month 12: number analyzed (Participants) | 3
  Month 12 | 2.0 (1.37)

4. Secondary Outcome: Coefficient of Variation of Glucose Value Per Each Subject Based on Continuous Glucose Monitoring Data
Description: The coefficient of variation of all available glucose value of each subject for each evaluation period is calculated, and then we present the mean and std of the individual coefficient of variation for each evaluation period.
Time Frame: Data is collected during the 7 days following the end of each period (At end of month 3, no glucose data is collected).
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Medtronic MiniMed Paradigm® REAL-Time System
Number analyzed (Participants) | 16
percentage
  Baseline: number analyzed (Participants) | 15
  Baseline | 36.3 (6.49)
  Month 6: number analyzed (Participants) | 12
  Month 6 | 30.5 (8.43)
  Month 9: number analyzed (Participants) | 6
  Month 9 | 31.0 (7.33)
  Month 12: number analyzed (Participants) | 3
  Month 12 | 24.3 (16.45)

5. Secondary Outcome: Mean Amplitude of Glycemic Excursion Based on Continuous Glucose Monitoring Data
Description: Mean Amplitude of Glycemic Excursion (which is often used to characterize glycemic variability, to know the detail of calculation, please refer to "Glucose Variability, © 2013 by the American Diabetes Association." ) of each subject for each evaluation period is calculated, and then we present the mean and std of the individual Mean Amplitude of Glycemic Excursion for each evaluation period.
Time Frame: Data is collected during the 7 days following the end of each period (At end of month 3, no glucose data is collected).
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Medtronic MiniMed Paradigm® REAL-Time System
Number analyzed (Participants) | 16
mmol/L
  Baseline: number analyzed (Participants) | 15
  Baseline | 6.9 (2.51)
  Month 6: number analyzed (Participants) | 11
  Month 6 | 6.8 (1.79)
  Month 9: number analyzed (Participants) | 6
  Month 9 | 6.7 (3.22)
  Month 12: number analyzed (Participants) | 2
  Month 12 | 5.5 (0.46)

6. Secondary Outcome: Number of Events in the Hypoglycemic Range
Description: Number of events in the hypoglycemic range (SG≤3.9mmol/L) of all available glucose value of each subject for each evaluation period is calculated, and then we present the mean and std of the individual number of events for each evaluation period.
Time Frame: Data is collected during the 7 days following the end of each period (At end of month 3, no glucose data is collected).
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: events
Arm/Group | Medtronic MiniMed Paradigm® REAL-Time System
Number analyzed (Participants) | 16
events
  Baseline SG≤3.9mmol/L: number analyzed (Participants) | 15
  Baseline SG≤3.9mmol/L | 0.5 (0.60)
  Month 6 SG≤3.9mmol/L: number analyzed (Participants) | 12
  Month 6 SG≤3.9mmol/L | 0.3 (0.54)
  Month 9 SG≤3.9mmol/L: number analyzed (Participants) | 6
  Month 9 SG≤3.9mmol/L | 0.1 (0.21)
  Month 12 SG≤3.9mmol/L: number analyzed (Participants) | 3
  Month 12 SG≤3.9mmol/L | 0.2 (0.17)

7. Secondary Outcome: Number of Events in the Hyperglycemic Range
Description: Number of Events in the Hyperglycemic Range (SG≥10.0 mmol/L) of all available glucose value of each subject for each evaluation period is calculated, and then we present the mean and std of the individual number of events for each evaluation period.
Time Frame: Data is collected during the 7 days following the end of each period (At end of month 3, no glucose data is collected).
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: events
Arm/Group | Medtronic MiniMed Paradigm® REAL-Time System
Number analyzed (Participants) | 16
events
  Baseline SG≥10.0 mmol/L: number analyzed (Participants) | 15
  Baseline SG≥10.0 mmol/L | 1.4 (0.73)
  Month 6 SG≥10.0 mmol/L: number analyzed (Participants) | 12
  Month 6 SG≥10.0 mmol/L | 1.4 (0.46)
  Month 9 SG≥10.0 mmol/L/L: number analyzed (Participants) | 6
  Month 9 SG≥10.0 mmol/L/L | 1.8 (0.83)
  Month 12 SG≥10.0 mmol/L: number analyzed (Participants) | 3
  Month 12 SG≥10.0 mmol/L | 1.1 (0.92)

8. Secondary Outcome: Area Under Curve in the Hypoglycemic Range
Description: Area under Curve in the hypoglycemic range (SG≤3.9mmol/L) of all available glucose value of each subject for each evaluation period is calculated, and then we present the mean and std of the individual Area under Curve for each evaluation period.
Time Frame: Data is collected during the 7 days following the end of each period (At end of month 3, no glucose data is collected).
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L*min
Arm/Group | Medtronic MiniMed Paradigm® REAL-Time System
Number analyzed (Participants) | 16
mmol/L*min
  Baseline SG≤3.9 mmol/L: number analyzed (Participants) | 15
  Baseline SG≤3.9 mmol/L | 0.03 (0.04)
  Month 6 SG≤3.9 mmol/L: number analyzed (Participants) | 12
  Month 6 SG≤3.9 mmol/L | 0.01 (0.03)
  Month 9 SG≤3.9 mmol/L: number analyzed (Participants) | 6
  Month 9 SG≤3.9 mmol/L | 0.00 (0.01)
  Month 12 SG≤3.9 mmol/L: number analyzed (Participants) | 3
  Month 12 SG≤3.9 mmol/L | 0.00 (0.00)

9. Secondary Outcome: Area Under Curve in the Hyperglycemic Range
Description: Area under Curve in the hyperglycemic range (SG≥10.0 mmol/L) based on all available glucose value of each subject for each evaluation period is calculated, and then we present the mean and std of the individual Area under Curve for each evaluation period.
Time Frame: Data is collected during the 7 days following the end of each period (At end of month 3, no glucose data is collected).
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L*min
Arm/Group | Medtronic MiniMed Paradigm® REAL-Time System
Number analyzed (Participants) | 16
mmol/L*min
  Baseline SG≥10.0 mmol/L: number analyzed (Participants) | 15
  Baseline SG≥10.0 mmol/L | 1.80 (1.55)
  Month 6 SG≥10.0 mmol/L: number analyzed (Participants) | 12
  Month 6 SG≥10.0 mmol/L | 1.94 (1.85)
  Month 9 SG≥10.0 mmol/L: number analyzed (Participants) | 6
  Month 9 SG≥10.0 mmol/L | 1.30 (1.36)
  Month 12 SG≥10.0 mmol/L: number analyzed (Participants) | 3
  Month 12 SG≥10.0 mmol/L | 0.32 (0.33)

10. Secondary Outcome: Percentage of Time in the Hypoglycemic Range
Description: Percentage of time in the hypoglycemic range (SG ≤ 3.9 mmol/L) of all available glucose value of each subject for each evaluation period is calculated, and then we present the mean and std of the individual percetage of time in that range for each evaluation period.
Time Frame: Data is collected during the 7 days following the end of each period (At end of month 3, no glucose data is collected).
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Medtronic MiniMed Paradigm® REAL-Time System
Number analyzed (Participants) | 16
percentage of time
  Baseline SG ≤ 3.9 mmol/L: number analyzed (Participants) | 15
  Baseline SG ≤ 3.9 mmol/L | 5.4 (6.87)
  Month 6 SG ≤ 3.9 mmol/L: number analyzed (Participants) | 12
  Month 6 SG ≤ 3.9 mmol/L | 1.8 (4.31)
  Month 9 SG ≤ 3.9 mmol/L: number analyzed (Participants) | 6
  Month 9 SG ≤ 3.9 mmol/L | 0.6 (1.26)
  Month 12 SG ≤ 3.9 mmol/L: number analyzed (Participants) | 3
  Month 12 SG ≤ 3.9 mmol/L | 0.6 (0.65)

11. Secondary Outcome: Percentage of Time in the Hyperglycemic Range
Description: Percentage of time in the hyperglycemic range (SG≥10.0 mmol/L) of all available glucose value of each subject for each evaluation period is calculated, and then we present the mean and std of the individual percentage of time in that range for each evaluation period.
Time Frame: Data is collected during the 7 days following the end of each period (At end of month 3, no glucose data is collected).
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Medtronic MiniMed Paradigm® REAL-Time System
Number analyzed (Participants) | 16
percentage of time
  Baseline SG ≥ 10.0 mmol/L: number analyzed (Participants) | 15
  Baseline SG ≥ 10.0 mmol/L | 44.1 (29.38)
  Month 6 SG ≥ 10.0 mmol/L: number analyzed (Participants) | 12
  Month 6 SG ≥ 10.0 mmol/L | 47.5 (32.87)
  Month 9 SG ≥ 10.0 mmol/L: number analyzed (Participants) | 6
  Month 9 SG ≥ 10.0 mmol/L | 36.6 (24.50)
  Month 12 SG ≥ 10.0 mmol/L: number analyzed (Participants) | 3
  Month 12 SG ≥ 10.0 mmol/L | 16.0 (14.77)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Medtronic MiniMed Paradigm® REAL-Time System
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 2/16
Other Adverse Events (participants affected / at risk) | 0/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medtronic MiniMed Paradigm® REAL-Time System (N=16)
Severe Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
hyperglycemia (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days